CLINICAL TRIAL: NCT01626781
Title: A Randomized, Open-label Phase III Trial of Mapisal® Versus an Urea Hand-foot Cream as Prophylaxis for Capecitabine-induced Hand-foot Syndrome in Patients With Gastrointestinal Tumors or Breast Cancer
Acronym: PROCAPP
Status: No longer available | Type: Expanded Access
Sponsor: AIO-Studien-gGmbH (Other)
Responsible Party: Sponsor
Other Study IDs: AIO-LQ-0111
Record Dates: First submitted 2012-06-21; First posted 2012-06-25 (Estimated); Last update posted 2013-10-22 (Estimated); Status verified 2013-10

CONDITIONS: the Treatment Hand-foot Syndrome Patients With Gastrointestinal Tumors or Breast Cancer, Who Are Treated With Capecitabine
MeSH Terms: conditions — Breast Neoplasms

INTERVENTIONS:
Device: Mapisal — Mapisal® ointment will be applied to hand and feet three times daily, as well as after washing hands. Treatment should start 2 days prior to the first chemotherapy cycle with capecitabine and will continue daily for the first 6 weeks of chemotherapy.
Other: Urea hand-foot cream — Urea hand-foot cream will be applied to hand and feet three times daily, as well as after washing hands. Treatment should start 2 days prior to the first chemotherapy cycle with capecitabine and will continue daily for the first 6 weeks of chemotherapy.

SUMMARY:
The purpose of this study is the examination of Mapisal® versus urea hand-foot cream as prophylaxis for capecitabine-induced hand-foot syndrome (HFS) in patients with gastrointestinal tumors or breast cancer, to assess the efficacy of Mapisal®.

Mapisal® is a medical device that is approved for the prophylaxis and treatment of HFS. Initial clinical data and case studies on the treatment and prophylaxis of Caelyx-induced HFS have been impressive. Because the pathomechanism of HFS caused by capecitabine is the same as for Caelyx-induced HFS, it is expected reason that administering Mapisal® should result in a significant reduction of HFS caused by capecitabine. The urea hand-foot cream was selected for the standard arm, because it is used commonly, is accepted by patients, and seems to have a positive influence on the severity of the HFS in the experience of many oncologists.

DETAILED DESCRIPTION:
Hand-foot syndrome (HFS) is a frequently occurring, often dose limiting, dermatologic reaction associated with cytotoxic agents, such as capecitabine, liposomal doxorubicin, and doxetacel.

Adverse events affecting the integument have posed significant challenges to oncologists in recent years in terms of selecting appropriate supportive therapies. Not only medications that inhibit EGFR receptors such as erlotinib, gefitinib, panitumumab or cetuximab, but also multiple-receptor tyrosine kinase inhibitors such as sunitinib and sorafenib and other "older" medications such as capecitabine can often lead to skin-related adverse events that can be difficult to manage.

These adverse events compromise skin-related quality of life and can lead to dose compromises or even the termination of treatment.

To date, there are no side effects reported for the use of either Mapisal® or urea hand-foot cream, making both treatments safe. Given the potential benefits of the treatments in preventing HFS by reducing discomfort and impairment of quality of life, the conduct of the trial is regarded as justifiable and there is no indication that patients are exposed to an increased risk associated with study participation.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. Male or female ≥18 years of age
3. Patients with gastrointestinal tumors or breast cancer who will be treated with capecitabine according to label
4. Palliative or adjuvant chemotherapy with capecitabine (combination- or mono-therapy, minimal dose of capecitabine 2000 mg/m2)
5. Life expectancy of least 12 weeks
6. WHO performance status 0-2
7. Adequate contraception
8. Willingness to fill in QoL forms
9. Laboratory requirements

   * Platelet count ≥100 × 109/L
   * Leukocyte count > 3.0 × 109/L
   * Hemoglobin ≥ 10.0 g/dL
10. Resolution of all chemotherapy- or radiotherapy-related toxicities to grade 1 or lower except for stable sensory neuropathy < grade 2. Any dermatological toxicities other than alopecia resulting from previous chemotherapy or radiotherapy must be completely resolved.

Exclusion Criteria:

1. Previous chemotherapy with capecitabine or liposomal doxorubicine, or any other substance, i.e. tyrosine kinase inhibitors (such as sorafenib and sunitinib) that may induce HFS
2. Radiotherapy or surgery within 4 weeks before start of treatment.
3. Dermatologic diseases that could interfere with the result of the clinical trial
4. Known drug/ alcohol abuse
5. Pregnant or breast feeding patients
6. Participation in another clinical trial and patient received investigational drug within the last 30 days prior to treatment start (i.e. follow-up within a preceding trial is not exclusionary)
7. Known allergic reactions to any of the ingredients of the ointments or capecitabine

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Deniz Gencer, Dr., Principal Investigator — Universitätsmedizin Mannheim
Locations (1):
- Universitätsmedizin Mannheim, III. Medizinische Klinik, Mannheim, Germany

REFERENCES:
- [Derived] Hofheinz RD, Gencer D, Schulz H, Stahl M, Hegewisch-Becker S, Loeffler LM, Kronawitter U, Bolz G, Potenberg J, Tauchert F, Al-Batran SE, Schneeweiss A. Mapisal Versus Urea Cream as Prophylaxis for Capecitabine-Associated Hand-Foot Syndrome: A Randomized Phase III Trial of the AIO Quality of Life Working Group. J Clin Oncol. 2015 Aug 1;33(22):2444-9. doi: 10.1200/JCO.2014.60.4587. Epub 2015 Jun 29. PMID 26124485
- See also: AIO - Working Group for Medical Onkology from the German Cancer Society — http://www.aio-portal.de